CLINICAL TRIAL: NCT02345083
Title: Indonesia Frailty, Aging, and Longitudinal Study
Acronym: INA-FRAGILE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Siti Setiati, Indonesia Frailty, Aging, and Quality of Life, Indonesia University
Other Study IDs: INA-FRAGILE01
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Frailty; Quality of Life
Keywords: Frailty; Pre-frailty; Fit; Robust; Elderly; Sociodemography status; Functional status; Cognitive status; Nutrition status; Comorbidity; Polypharmacy; Mortality; Depression status; Health-related quality of life; Fall incidence; Hospitality
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Frailty is a dynamic process from fit (robust) and pre-frail elderly. There is no previous study that determine the risk factors from fit to pre-frailty and pre-frailty to frailty in Indonesian elderly.

This study was aimed to define the risk factors and clinical outcomes of frailty transitional status in Indonesian elderly.

DETAILED DESCRIPTION:
Frailty is an age-associated, biological syndrome characterized by decreased biological reserves, due to dysregulation of several physiological systems, which puts an individual at risk when facing minor stressors, and is associated with poor outcomes (ie, disability, death, and hospitalization).

Frailty identifies a high-risk subgroup and offers characteristics of great clinical importance: a higher reversibility at early stages than disability, and a higher predictive value than chronic disease for adverse outcomes at older ages. It is also the most common condition leading to death in community-dwelling older people.

However, there is current consensus that physical frailty is potentially reversible. It is hence useful to objectively detect frailty among frail elderly persons, as frailty indices serve a useful purpose for risk stratification, predicting need for institutional care and planning of services needed.

To date, there is no study or information about frailty status in Indonesia elderly. This study was aimed to define the risk factors and clinical outcomes of frailty transitional status in Indonesian elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly aged >= 60 years old
2. Fit (robust) or pre-frailty;
3. Capable to understand and carry-out the instruction.

Exclusion Criteria:

1. Unwilling to join the study;
2. Abbreviated Mental Test (AMT) score < 8;
3. Geriatric Depression Scale (GDS) score >= 10;
4. Body mass index (BMI) <18,5 Kg/m2;
5. Malnutrition (according to Mini Nutritional Assessment/MNA);
6. Liver cirrhosis, severe liver dysfunction, or serum ALT levels >3 times upper normal limit;
7. Acute illness during inclusion period, eg. pneumonia, pain due to acute arthritis (visual analog scale >6/10), stroke attack, crisis hypertension;
8. Severe cardiac dysfunction: acute decompensated heart failure and/or chronic heart failure functional class III or IV (New York Heart Association classification);
9. Severe pulmonary dysfunction: acute exacerbation of chronic obstructive lung disease stage III or IV (GOLD classification), and/or PaO2 levels < 60 mmHg.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fit or pre-frail elderly aged >= 60 years old who came to Comprehensive Geriatric Clinics, Cipto Mangunkusumo General Hospital, Jakarta, during March 2015-March 2016.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in frailty status at 1 year | Baseline and at 1 year
  Frailty status is divided into Fit (robust), Pre-frail, and Frailty.

SECONDARY OUTCOMES:
Change from baseline in health-related quality of life at 1 year | Baseline and at 1 year
  Health-related quality of life: using Euro Quality of Life-5 Dimension (EQ-5D) questionnaire.
Change from baseline in fall incidence at 1 year | Baseline and at 1 year
  Fall incidence: number of fall during observational period.
Change from baseline in hospitality at 1 year | Baseline and at 1 year
  Hospitality: number of hospital admission (emergency or inpatient care) during observational period.
Change from baseline in mortality at 1 year | Baseline and at 1 year
  Mortality: number of subjects died after 1 year observation.

OTHER OUTCOMES:
Change from baseline in handgrip strength at 1 year | Baseline and at 1 year
  Measurement: using Jamar Hydraulic Hand Dynamometer Model J00105
Change from baseline in gait speed at 1 year | Baseline and at 1 year
  Measurement: 15-feet walking test
Change from baseline in functional status at 1 year | Baseline and at 1 year
  Measurement: Barthel Index Activities of Daily Living (B-ADL) & Lawton Instrumental & Activities of Daily Living (L-IADL) questionnaires.
Change from baseline in cognitive status at 1 year | Baseline and at 1 year
  Measurement: Abbreviated mental test (AMT) questionnaire.
Change from baseline in mental status at 1 year | Baseline and at 1 year
  Measurement: Short Form Geriatric Depression Scale (GDS) questionnaire.
Change from baseline in nutritional status at 1 year | Baseline and at 1 year
  Measurement: Mini Nutritional Assessment (MNA) questionnaire.
Change from baseline in sarcopenia status at 1 year | Baseline and at 1 year
  Categories: no sarcopenia, pre-sarcopenia, sarcopenia, and severe sarcopenia.
Change from baseline in comorbidities status at 1 year | Baseline and at 1 year
  Measurement: Cumulative Illness Rating Scale (CIRS)

CONTACTS AND LOCATIONS:
Overall Officials: Siti Setiati, Prof, MD, Principal Investigator — Division of Geriatrics, Department of Internal Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta; Purwita Laksmi, MD, Study Chair — Division of Geriatrics, Department of Internal Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta; Tirza Tamin, MD, PhD, Study Chair — Department of Rehabilitation & Physical Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta; Rahmi Istanti, SKM, MARS, Study Chair — Division of Geriatrics, Department of Internal Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta
Locations (1):
- Comprehensive Geriatric Clinic, Cipto Mangunkusumo Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Lee JS, Auyeung TW, Leung J, Kwok T, Woo J. Transitions in frailty states among community-living older adults and their associated factors. J Am Med Dir Assoc. 2014 Apr;15(4):281-6. doi: 10.1016/j.jamda.2013.12.002. Epub 2014 Feb 16. PMID 24534517
- [Background] Laksmi PW. Frailty syndrome: an emerging geriatric syndrome calling for its potential intervention. Acta Med Indones. 2014 Jul;46(3):173-4. No abstract available. PMID 25348178